CLINICAL TRIAL: NCT03094637
Title: A Phase II Study of the Combination of Azacitidine and Pembrolizumab for Patients With MDS
Brief Title: Azacitidine and Pembrolizumab in Treating Patients With Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0343; NCI-2018-01238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0343 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Results first posted 2021-10-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: High Risk Myelodysplastic Syndrome; IPSS Risk Category Intermediate-1; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, pembrolizumab) (Experimental): Patients receive azacitidine Intravenous (IV) over 10-40 minutes or Subcutaneous (SC) on days 1-7, and pembrolizumab IV over 30 minutes every 3 weeks. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the side effects of azacitidine and pembrolizumab and to see how well they work in treating patients with myelodysplastic syndrome. Azacitidine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving azacitidine and pembrolizumab may work better at treating myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of the combination of azacitidine and MK3475 (pembrolizumab) in patients with higher risk myelodysplastic syndrome (MDS).

II. To explore the clinical activity (response, survival effect) of the combination of azacitidine with MK-3475 in patients with higher risk MDS.

EXPLORATORY OBJECTIVES:

I. To study the biological effects of the combination of azacitidine and pembrolizumab in patients with MDS treated on this study.

OUTLINE:

Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1-7, and pembrolizumab IV over 30 minutes every 3 weeks. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days, every 12 weeks for 1 year, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signed informed consent before performance of any study related procedure not part of normal medical care indicating that the patient is aware of the investigation and nature of this study in keeping with institutional policies and with the understanding that the consent may be withdrawn with the subject at any time without prejudice to future medical care
* Intermediate 1 (INT-1) or higher risk MDS defined by International Prognostic Scoring System (IPSS) criteria
* Patients can or cannot have receive prior therapy with hypomethylating agent but will be allocated to specific patient cohorts based on their prior exposure. Patients that had received prior hypomethylating agent therapy should have at least received 6 cycles of therapy and not achieved any response or had progressed after any given number of cycles
* Eastern Cooperative Oncology Group (ECOG) performance of 0 to 2
* Male patients, even if surgically sterilized, should agree to practice effective barrier contraception for the entire study treatment period and through 120 days after the last dose of the study treatment or agree to completely abstain from heterosexual intercourse. Female patients who are postmenopausal for at least one year before the screening visit or are surgical sterile or if they are of child bearing potential must have a negative pregnancy test within 72 hours of treatment of the start date and agree to practice two effective methods of contraception forms at the same time from the time of signing the informed consent through 120 days of the last dose of the study treatment or agree to completely abstain from heterosexual intercourse
* Willingness and ability to comply with scheduled visits treatment plans, laboratory tests and other study procedures
* Serum creatinine or measured or calculated creatine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrcL]) =< 2.0 x upper limit of normal (ULN) or >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (performed within 10 days of treatment initiation). Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 2.0 x ULN (unless considered due to Gilbert's disease or leukemia disease) or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (unless considered due to Gilbert's disease or leukemia disease) or =< 5 x ULN for subjects with liver metastases (performed within 10 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Patients must receive a minimum dose of azacitidine of 75mg/(m)(2) dose

Exclusion Criteria:

* Significant medical psychiatric cognitive or other conditions that may compromise the patient ability to understand the patient information to give informed consent to comply with the study protocol or to complete the study
* Any severe or concurrent disease or condition including uncontrolled systemic infection, congestive heart failure, angina pectoris or cardiac arrhythmia and autoimmune processes that in the opinion of the investigator would make the patient inappropriate for study participation
* Patients with known hypersensitivity to 5-azacitidine or MK3475 or any of their excipients
* Prior history of stem cell transplantation
* For patients in the relapse or refractory cohort, any other therapy not being a hypomethylating agent after hypomethylating agents (HMA) failure or more than 4 months since completion of last cycle of hypomethylating agent. Please note that hypomethylating agent may include second generation compounds such as SGI-110, oral decitabine or oral azacitidine and will also include combinations with investigational agents
* Treatment with other investigational agents including chemotherapy, immunotherapy, or radiation therapy within a month prior to the start of this clinical trial
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2023-11-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2017 to March 2020
Groups:
- Treatment (Azacitidine, Pembrolizumab) in Untreated Patients; Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) failureHMA Failure: Patients receive azacitidine IV over 10-40 minutes or SC on days 1-7, and pembrolizumab IV over 30 minutes every 3 weeks. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given IV
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) failureHMA Failure
Started | 17 | 20
Completed | 17 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) Failure: Patients receive azacitidine IV over 10-40 minutes or SC on days 1-7, and pembrolizumab IV over 30 minutes every 3 weeks. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Azacitidine: Given IV
  Pembrolizumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) Failure | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 13 | 20 | 33
Age, Continuous [Median (Full Range); unit: years] | 72 [36 to 83] | 75 [65 to 84] | 74 [36 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 10 | 15 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Defined as Complete Response + Partial Response + Hematological Improvement
Description: Will estimate the ORR for the experimental treatments, along with the 95% credible intervals. The association between ORR and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Time Frame: Up to 2 years 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) Failure
Number analyzed (Participants) | 17 | 20
Participants | 13 | 5

2. Primary Outcome: Event Free Survival
Description: Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) failureHMA Failure
Number analyzed (Participants) | 17 | 20
Months | 9.24 [3.98 to 31.23] | 5.39 [1.48 to 9.07]

3. Primary Outcome: Overall Survival
Description: Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests. Overall Survival will be presented by median survival, which is the time point at which the cumulative survival drops below 50%. If there is no median survival (not reached), it means the cumulative survival was more than 50%.
Time Frame: Up to 4 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) failureHMA Failure
Number analyzed (Participants) | 17 | 20
Months | NA [1 to 32] — Median survival for frontline patients cohort was not reached as the cumulative survival was greater than 50%. | 5.79 [4.47 to 18.61]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) Failure
All-Cause Mortality (participants affected / at risk) | 1/17 | 2/20
Serious Adverse Events (participants affected / at risk) | 9/17 | 13/20
Other Adverse Events (participants affected / at risk) | 15/17 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients (N=17) | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) Failure (N=20)
Hyperbilirubinemia (Investigations) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 1 (1) | 2 (4)
fever (General disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 4 (6) | 11 (12)
Infection G 3 or 4 neutrophils (Infections and infestations) | 1 (1) | 1 (1)
Intra-operative Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal/Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Azacitidine, Pembrolizumab) in Untreated Patients (N=17) | Treatment (Azacitidine, Pembrolizumab) Patients With Hypomethylating Agent (HMA) Failure (N=20)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Alanine Aminotransferase (Investigations) | 1 (1) | 4 (4)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asparatate Aminotransferase (Investigations) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (6)
Dermatology Skin/Other (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2)
anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 1 (2)
Injection Site Reaction (General disorders) | 1 (1) | 2 (2)
Neutropenia (Investigations) | 3 (3) | 7 (7)
Pain (General disorders) | 6 (6) | 3 (3)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03094637/Prot_SAP_000.pdf